CLINICAL TRIAL: NCT06898775
Title: Retrospective Analysis of Passive Safety Surveillance Data of Dengue Vaccine, Qdenga (TAK 003) At Private Vaccination Centers, During 2023 and 2024 Dengue Season in Buenos Aires, Argentina
Brief Title: Passive Safety Surveillance Data of Dengue Vaccine, Qdenga (TAK 003) in Private Vaccination Sites in Buenos Aires, Argentina.
Status: Active, not recruiting | Type: Observational
Sponsor: Fundación Vacunar (Other)
Responsible Party: Sponsor
Other Study IDs: Fundación Vacunar
Record Dates: First submitted 2025-03-21; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Dengue Vaccines
Keywords: Dengue; vaccine; safety; passive surveillance; AEFI; TAK-003; Argentina
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Individuals vaccinated with Qdenga at Vacunar centers since November 2023- Nov 2024: Participants from 4 years of age with no upper limit in accordance with ANMAT approval and for whom safety data is available through the Vacunar centers passive surveillance systems

SUMMARY:
The TAK-003 vaccine, Qdenga, developed by Takeda, was approved by ANMAT in April 2023 and has been available in Argentina since November 2023 for individuals from 4 years old and without limit of age. Clinical trials demonstrate that Qdenga has a favorable safety profile, adequate immunogenicity for all four serotypes, and efficacy in preventing severe dengue in seropositive and seronegative subjects. However, there are currently limited real-world safety studies on TAK-003, particularly for adults over 60 years old.

The aim of this study is to evaluate Adverse Events Supposedly Attributed to Vaccination and Immunization (AEFI) for TAK-003 vaccine in vaccinated people at private vaccination centers in Buenos Aires metropolitan area.

ELIGIBILITY:
Inclusion Criteria:

* All individuals who were vaccinated with Qdenga at Vacunar centers since November 2023 still 1st November 2024, from 4 years of age with no upper limit in accordance with ANMAT approval and for whom safety data is available through the Vacunar centers passive surveillance systems.

Exclusion Criteria:

* Reports with insufficient information to characterize the AEFI will be excluded from the analysis.

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: People vaccinated with dengue vaccine, TAK-003 at private vaccination centers in Buenos Aires, Argentina
Sampling Method: Non-Probability Sample
Enrollment: 112345 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEFI | 42 days
  The incidence of AEFI will be calculated in terms of the number of notifications per 1,000 doses administered.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación Vacunar, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided